CLINICAL TRIAL: NCT03900260
Title: Clinical Evaluation of the Lenstec Softec HP1 Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lenstec Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR505
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Aphakia
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Softec HP1 Intraocular Lens (Other): The Softec HP1 IOL is a single-piece, biconvex, ultraviolet absorbing intraocular lens designed for insertion into the posterior chamber of the human eye for visual correction of Aphakia in adults over the age of 21, and as a replacement of a damaged (cataract) natural lens.
  Interventions: Device: Softec HP1 Intraocular Lens

INTERVENTIONS:
Device: Softec HP1 Intraocular Lens — The Softec HP1 IOL is a single-piece, biconvex, ultraviolet absorbing intraocular lens designed for insertion into the posterior chamber of the human eye for visual correction of Aphakia in adults over the age of 21, and as a replacement of a damaged (cataract) natural lens.

SUMMARY:
The study is designed as a post market evaluation of the Softec HP1 IOL for continuance of the CE certificate. The primary effectiveness endpoint is to evaluate the safety and performance levels produced by this IOL in patients requiring standard cataract surgery. There will be no change from standard procedure, other than 1 extra post op evaluation.

DETAILED DESCRIPTION:
Recruitment will be performed by the 3 Clinical Investigators (Jean-Pierre Danjoux - Sunderland Eye Infirmary, Karen Goodall - Croft Shifa Health Center, Mark Benson - Midland Eye Institute) and any appropriate, pre-trained staff within the hospital using the inclusion and exclusion criteria set out in the protocol. Patient selection will involve anyone over the age of 21 with an age-related cataract regardless of ethnicity, religion or gender.

An Informed Consent Form (ICF) will be explained with patients in full which will be signed by both the Principal Investigator (PI) and the patient with full understanding. Understanding fully means that the patient understands the nature of the operation, the benefits to the operation and also any risks or burdens.

The consent form also states alternatives to participation in the trial other than the option being put forward. The patients will be of sound enough mind to retain the information from the ICF and will be given time to digest this in order to make a free and effective decision to join the study.

All risks and benefits are explained in the ICF and are no more or less than that of a standard cataract surgery provided on a daily basis by NHS consultants. All surgeries will be performed by the PI.

Confidentiality shall be kept at all times with the PI and clinical staff using a unique patient reference number that in no instance indicates the identity of the patient to the study sponsor (Lenstec Inc.) or anyone else outside of the hospital. Any other confidentiality issues will run in conjunction with the hospital policy of which the staff involved in the study are aware.

There are no tissue samples to be used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 21 years of age, of any race and either gender
2. Operable, age related cataract grade in one or both eyes
3. Patients who require an IOL power in the range of 10.0 - 30.0 D only
4. Able to comprehend and sign a statement of informed consent
5. Planned cataract removal by phacoemulsification
6. Potential postoperative visual acuity of 0.2 logMAR or better
7. No other ocular or systemic pathology that may affect visual outcome following cataract surgery
8. Clear intraocular media other than cataract in study eyes
9. Preoperative Best Corrected Visual Acuity (BCVA - VA taken with original manifest refraction) worse than 0.2 logMAR
10. Able to competently complete testing
11. Willing and able to attend study visits

Exclusion Criteria:

1. Previous intraocular surgery
2. Previous corneal refractive surgery
3. Any inflammation or oedema (swelling) of the cornea
4. Pterygium with corneal involvement or has the potential of corneal involvement (in the opinion of the Investigator)
5. Amblyopia
6. Clinically significant ptosis
7. Clinically severe corneal dystrophy (e.g. epithelial, stromal, or endothelial dystrophy), keratitis, keratoconjunctivitis, keratouveitis, keratopathy, or kerectasia
8. Diabetic Retinopathy
9. Previous retinal detachment
10. Previous corneal transplant
11. Iris neovascularization
12. Glaucoma (medically controlled or uncontrolled)
13. Aniridia
14. Chronic severe uveitis
15. Optic nerve atrophy
16. Corneal decompensation
17. History of corneal disease (e.g. herpes simplex, herpes zoster keratitis, etc.)
18. Pseudoexfoliation syndrome
19. Iris atrophy
20. Aniseikonia
21. Pregnant, lactating, or planning to become pregnant during the course of the trial Note: Patients who become pregnant during the study will not be discontinued; however, data may be excluded from the effectiveness analyses because pregnancy can alter refraction and visual acuity results.
22. Participation in another clinical trial within 30 days of study start

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Best Corrected Distance Visual Acuity (BCDVA) | 3 months
  The postoperative BCDVA for up to 75 patients will be measured under normal lighting conditions using a phoropter or trial frames, and these results will be evaluated by the sponsor on completion of the study.

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UCDVA) | 3 months
  The postoperative UCDVA for up to 75 patients will be measured under normal lighting conditions using a phoropter or trial frames, and these results will be evaluated by the sponsor on completion of the study.

OTHER OUTCOMES:
Complication Rates | 3 months
  Up to 75 patients will be evaluated for intraoperative and postoperative complications, and these will be compared to the complication rates provided in the FDA Grid.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Danjoux, MD, Principal Investigator — Sunderland Eye Infirmary; Karen Goodall, MD, Principal Investigator — Croft Shifa Health Center; Mark Benson, MD, Principal Investigator — Midland Eye Institute
Locations (3):
- United Kingdom (3):
  - Croft Shifa health Centre, Rochdale
  - Midland Eye Institute, Solihull
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No